CLINICAL TRIAL: NCT01537172
Title: A Phase 1, Single Centre, Three-part, Randomised, Study to Investigate the Safety, Tolerability and Pharmacokinetic Profile of Single and Multiple Ascending Doses of Oral ONO-4053 and the Effects of Food in Healthy Males and Females
Brief Title: A Phase I Study to Evaluate Safety, Tolerability and Pharmacokinetics of ONO-4053 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-4053POE002
Record Dates: First submitted 2012-02-13; First posted 2012-02-23 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Adult Subjects
Keywords: ONO-4053 healthy subjects; 3 part adaptive design

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ONO-4053 (Experimental): E Experimental Intervention Drug: ONO-4053
  Interventions: Drug: ONO-4053
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-4053 — Part A: ONO-4053 doses proposed are 10 mg, 30 mg, 100 mg, 300 mg, 600 mg, 900 mg as a single dose administered by mouth once daily, depending on the outcome of the previous dose.
  Arms: ONO-4053
Drug: Placebo — Placebo to match ONO-4053 tablets, dosed in a similar manner to ONO-4053
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of ONO-4053 across ascending single and multiple doses in healthy adult male and female subjects.

The secondary objective of the study is to characterize the pharmacokinetic profile of ONO-4053 in healthy adult male and female subjects.

DETAILED DESCRIPTION:
Ono Pharma UK Ltd is the European subsidiary of Ono Pharmaceutical Co. Ltd. As the European Legal Representative of Ono Pharmaceutical Co. Ltd, Ono Pharma UK Ltd is carrying out this study.

This is a clinical study of ONO-4053 in healthy volunteers. This study consists of three parts. Part A will investigate the safety, tolerability and pharmacokinetics when single ascending doses of ONO-4053 are administered in a double-blind manner. Part B will investigate the pharmacokinetics of ONO-4053 in the fed and fasted state in an open-label manner. Part C will investigate the safety, tolerability and pharmacokinetics when multiple ascending doses of ONO-4053 are administered in a double-blind manner. Doses for Part B and C will be determined after data from Part A are available.

ELIGIBILITY:
Inclusion Criteria:

* Healthy caucasian subjects aged 18-45 years inclusive.
* Subjects with a body mass index of 19-30 kg/m2 inclusive and who weigh at least 50 kg and no more than 100 kg at screening.

Exclusion Criteria:

* Subjects who have a clinically relevant history or presence of any clinically significant disease or disorder.
* Current smokers or those that have smoked or used nicotine products within 6 months of the Screening visit.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ONO-4053 across ascending single and multiple doses using adverse events, vital signs, 12-lead ECG, continuous ECG monitoring and clinical lab tests. | Day 17

SECONDARY OUTCOMES:
Plasma and urine concentrations of ONO-4053 and derived pharmacokinetic parameters | Day 17

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Department, Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Hammersmith Medicines Research Ltd, London, United Kingdom